CLINICAL TRIAL: NCT03926897
Title: Blood Pressure Measuring Practice of Hong Kong Primary Care Doctors: a Cross-sectional Study
Brief Title: Blood Pressure Measuring Practice of Hong Kong Primary Care Doctors
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: SBRE-18-563
Record Dates: First submitted 2019-04-19; First posted 2019-04-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: While office BP measurements were traditionally used to detect, diagnose and manage hypertension(HT), studies had convincingly showed that out-of-office blood pressure, including home blood pressure monitoring (HBPM) and ambulatory blood pressure monitoring (ABPM), was superior in predicting cardiovascular outcomes and death. Furthermore, some countries' guidelines suggested the use of validated automatic blood pressure machines (called automated office blood pressure monitoring (AOBP)) to screen for HT and record BP in routine HT clinical management. With difference between guidelines and various available BP measurement methods, it is not known how primary care doctors, who play the key role to detect and treat HT, are measuring BP in their daily practice.

Method: All doctors registered in the primary care directory will be mailed a questionnaire. Those who do not respond would be mailing for maximally 3 times, 2 weeks apart to enhance response rate. It is estimated that around 1500-2000 doctors will be eligible.

ELIGIBILITY:
Inclusion Criteria:

* All doctors registered in the primary care directory in Hong Kong

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctors who regarded themselves working in Primary Care in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
the blood pressure (BP) measurement method for screening of hypertension | 1 year
  possible answers included: Manual BP in the office with mercury or aneroid device; Manual BP in the office with an electronic device; Automated office BP machines (AOBP) ; Other patient-activated electronic devices in the office; Electronic BP kiosks
The BP measurement method to diagnose hypertension | 1 year
  possible answers included: Manual BP in the office with mercury or aneroid device; Manual BP in the office with an electronic device; Automated office BP machines (AOBP) ; Other patient-activated electronic devices in the office; Electronic BP kiosks; Ambulatory BP monitoring (24-hour to 48-hour BP monitoring); home BP monitoring
your routine methods used to measure BP in patients taking antihypertensive treatment (lifestyle or medications) | 1 year
  possible answers included: Manual BP in the office with mercury or aneroid device; Manual BP in the office with an electronic device; Automated office BP machines (AOBP) ; Other patient-activated electronic devices in the office; Electronic BP kiosks; Ambulatory BP monitoring (24-hour to 48-hour BP monitoring); home BP monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
will share information when required by other researchers

REFERENCES:
- [Derived] Lee EKP, Choi RCM, Liu L, Gao T, Yip BHK, Wong SYS. Preference of blood pressure measurement methods by primary care doctors in Hong Kong: a cross-sectional survey. BMC Fam Pract. 2020 May 26;21(1):95. doi: 10.1186/s12875-020-01153-6. PMID 32456619